CLINICAL TRIAL: NCT00160849
Title: Study on the Feasibility of Antiretroviral Therapy With a Single Agent - Lopinavir/r - in Patients Treated With HAART and With Viral Load Below 80 Copies/Ml
Brief Title: Lopinavir/r Monotherapy as Maintenance Therapy After Long Term Viral Suppression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KalMo
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Lopinavir/r

SUMMARY:
1. Objectives Primary

   * To investigate the possibility of maintaining virological suppression of HIV in infected patients, switching them to LPV/r as the only antiretroviral agent
   * To assess the immunological response in patients who switched to LPV/r as single agent, based on the observation of changes in the serum levels of CD4+ cells.

   Secondary
   * To investigate the rate of clinical and laboratorial adverse events in the two treatment groups.
   * To investigate the rate of emergence of antiretroviral resistance mutations in the two treatment groups, in case of virological failure of the current regimen.
   * To describe the adherence to the prescribed regimen in the two treatment groups
   * To describe changes in body fat distribution (abdominal, arms and thigh circumference) and in the lipid profile, in patients from the two treatment groups
   * To describe the rate of clinical failure of the antiretroviral therapy in the two treatment groups.
2. Patient population:

   The 60 patients were selected by the investigators according to the study's inclusion and exclusion criteria, and were divided into 2 groups with 30 patients each.
3. Study design:

   The study is multicentric, open-label, randomized. Virological, immunological and clinical failures will be analyzed in both groups. In addition, data on clinical or laboratorial toxicity and compliance are being recorded.
4. Regime:

   * Group 1 maintenance of the currently used antiretroviral therapy
   * Group 2 switch to LPV/r antiretroviral monotherapy in the dose of 400/100 mg 12/12 hs with food. Patients in group 2 who were being treated previously with non-nucleoside reverse transcriptase inhibitors (Efavirenz or Nevirapine) were instructed to take 4 capsules of Lopinavir/r each 12 hs, during the first 14 days of therapy (up to Week 2 visit).
5. Duration:

96 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

1. The patients must fulfill all of the following criteria: The patient has confirmed his/her willingness to participate in the study, after being informed about all the aspects of the study that might be relevant for his/her decision to participate, and has signed and dated the informed consent form, as approved by the Institutional Review Board/ Ethics Committee (IRB/EC). And he/she can withdraw the study participation at any moment, if he/she wants to do so.
2. The patient has laboratorial confirmation of an HIV infection through a positive ELISA test for anti-HIV antibodies and an additional test (Western-blot, indirect immunofluorescence or PCR).
3. The patient must be in treatment with at least three antiretroviral drugs, for at least 6 months without changes.
4. The patient should have no history of documented virological failure to previously used antiretroviral therapies.
5. Undetectable viral load (test result < 400 copies/ml) for more than 6 months measured on a sample collected during treatment with the current regimen and at screening (test result < 80 copies).
6. CD4 count > 200 cels/ml at screening
7. Patient agrees not to use concomitant medication that might have unacceptable drug interactions with the study drug.
8. If the patient is a female, she must have a negative pregnancy test and must agree to use at least 14 days before the study drug administration and for the whole study duration and up to 6 months after, a barrier contraceptive method with a proven reliability track record, as judged by the investigator

Exclusion Criteria:

1. Pregnant or lactating female patient. If the patient becomes pregnant during the study, she will be discontinued from the study.
2. Patients with allergic reaction or hypersensitivity to Lopinavir or Ritonavir .
3. A patient with previous history of opportunistic disease ( appendix 1) or CD4 count below 100 cels/mm3.
4. A patient who presents any HIV viral load test result above 400 copies/mL over the past 6 months.
5. Patient who is receiving or has received systemic chemotherapy during the past 6 months.
6. Laboratory test results Hemoglobin < 8 g/dl Absolute neutrophil count < 750 cels/mL Platelet count < 20,000/mL Bilirubin > 1.5 x UNL or > 6 x UNL if patient is using Indinavir or Atazanavir ALT and AST > 2 x UNL Creatinine > 2 x UNL
7. Patient is taking any drug known to be contraindicated concomitantly with lopinavir/r. Please refer to the product's package insert.
8. According to the investigator's opinion, the patient has little probability of complying with the study protocol or is unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2007-03

PRIMARY OUTCOMES:
• Rate of suppression of viral load to less than 80 copies/ml on weeks 4, 12, 24, 36, 48, 60, 72, 84, 96.
• Average change of CD4 count on weeks 4, 12, 24, 36, 48, 60, 72, 84, 96
• Two-year incidence rate of immunodeficiency related clinical conditions.

SECONDARY OUTCOMES:
• Toxicity rate (clinical and laboratorial adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: Estevão P Nunes, M.Sc, Principal Investigator — Projeto Praça Onze
Locations (2):
- Brazil (2):
  - Hospital Geral de Nova Iguaçu, Nova Iguaçu, Rio de Janeiro
  - Projeto Praça Onze, Rio de Janeiro, Rio de Janeiro